CLINICAL TRIAL: NCT04967209
Title: Investigation of a Digital Healthy Habits Program for Individuals With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Noom Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 00055029
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Breast Cancer; Obesity; Overweight and Obesity; Overweight
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This mixed methods study will involve obtaining user feedback on the first 4 weeks of the Healthy Habits for Cancer (HCC) Program. Short pre and post surveys and in-depth qualitative interviews will be conducted exploring their views on the app (features they liked and didn't like), the extent to which they believe the app would have to be further adapted, how they would feel about such an app being embedded in their cancer care and when in their care pathway they would like to be offered it.

DETAILED DESCRIPTION:
This mixed methods study will involve obtaining user feedback on the first 4 weeks of the Healthy Habits for Cancer (HCC) Program. Participants will be recruited and asked to try the HCC app for 4 weeks. Short pre and post surveys and in-depth qualitative interviews will be conducted exploring their views on the app, the extent to which they believe the app would have to be further adapted, how they would feel about such an app being embedded in their cancer care and when in their care pathway they would like to be offered it.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* 18 years and older
* Female
* > 6 months postpartum
* Not currently pregnant or planning to become pregnant in the next 5 months
* Diagnosed with stage I-IV breast cancer < 5 years ago:
* Completed active breast cancer treatment (e.g., chemotherapy, radiation, surgery) 1 month to 5 years ago, with the exception of hormonal/endocrine therapy
* Currently prescribed hormone therapy (e.g. Tamoxifen) as a breast cancer treatment
* Not diagnosed with an eating disorder
* Healthy weight, overweight, or obesity (BMI ≥ 18.5)
* Willingness to use the program over the course of the 4 weeks in order to enable them to provide feedback on its features
* Own a smartphone with iOS operating system (i.e., Apple iPhone)

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent
* Underweight (BMI < 18.5)
* Currently pregnant or <6 months postpartum
* Presence of a diagnosed physical or mental health condition or abnormality that impacts the ability to participate in a program that involves asking participants to monitor diet, physical activity, or weight (e.g., eating disorder, bipolar disorder). If there is any doubt at initial screening the investigator will recommend that the patient receives sign off from their clinical team.
* Currently undergoing IV chemotherapy or radiation
* Plans for surgery in the next 6 weeks
* Currently diagnosed or being treated for a second primary cancer (i.e. cancer of another organ, not due to breast cancer metastasis), with the exception of non-melanoma skin cancers (e.g. basal cell carcinoma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with breast cancer diagnosis currently undergoing hormone therapy for treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast quality-of-life instrument | 4 weeks
  Self reported measure of multidimensional quality of life (QL) in patients with breast cancer.
Qualitative interviews | 4 weeks
  Data analyses will content analyze key themes in participants' experiences using the program, including their likes and dislikes for the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Noom, Inc, New York, New York, United States